CLINICAL TRIAL: NCT00887276
Title: Prospective, Doubleblind, Randomized Multicenter Study to Proof the Clinical and Bacteriological Non-inferiority of Ampicillin/Amoxicillin Versus Moxifloxacin in Hospitalized Patients With Non-severe Community-acquired Pneumonia
Brief Title: Study to Proof the Clinical and Bacteriological Non-inferiority of Ampicillin/Amoxicillin Versus Moxifloxacin in Hospitalized Patients With Non-severe Community-acquired Pneumonia
Acronym: PENCAP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: CAPNETZ Stiftung (Other)
Responsible Party: Prof. Dr. Reinhard Marre, University of Ulm
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT number: 2005-000771-18
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2010-01

CONDITIONS: Community Acquired Pneumonia
Keywords: Ampicillin; Amoxicillin; Moxifloxacin; Community-Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin
- Ampicillin; Amoxicillin (Active Comparator)
  Interventions: Drug: Ampicillin;Amoxicillin

INTERVENTIONS:
Drug: Moxifloxacin — intravenous infusion: at least 3 days until to the drug switch (oral use),3 times daily (all 8 hours)
  1. 20 ml physiologic saline solution (placebo)(over 30 min) + Moxifloxacin infusion solution(400 mg/250ml) over 60 minutes
  2. 20 ml physiologic saline solution (placebo) (over 30 min)
  3. 20 ml physiologic saline solution (placebo) (over 30 min)
  following oral therapy(possible at the earliest day 4): 3 times daily (all 8 hours):
  1. 1 capsule Moxifloxacin (400 mg) + 1 capsule Placebo
  2. 2 capsules Placebo
  3. 2 capsules Placebo
  Total time of the therapy:at least 7 days, but at most 10 days
  Other Names: Avalox
  Arms: Moxifloxacin
Drug: Ampicillin;Amoxicillin — intravenous infusion:at least 3 days until to the drug switch (oral use), 3 times daily (all 8 hours)
  1. 2 g Ampicillin dissolved in 20 ml aqua (i.v. over 30 min) + 250 ml physiologic saline solution (placebo) (over 60 min)
  2. 2 g Ampicillin dissolved in 20 ml aqua (i.v. over 30 min)
  3. 2 g Ampicillin dissolved in 20 ml aqua (i.v. over 30 min)
  following oral therapy(possible at the earliest day 4): 3 times daily (all 8 hours):
  1. 2 capsules Amoxicillin (0,5 g)
  2. 2 capsules Amoxicillin (0,5 g)
  3. 2 capsules Amoxicillin (0,5 g)
  Total time of the therapy: at least 7 days, but at most 10 days
  Other Names: Ampicillin Ratiopharm; Amoxicillin ratiopharm
  Arms: Ampicillin; Amoxicillin

SUMMARY:
The purpose of this study is to prove the clinical and bacteriological non-inferiority of ampicillin/amoxicillin versus moxifloxacin in hospitalized patients with non-severe community-acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Men or women older than 18 years with signed informed consent
* Women in a childbearing age with sufficient conception protection or if necessary negative pregnancy test
* Infiltrates appeared newly in the x-ray thorax
* Breath-conditioned chest pain
* At least two of the following clinical symptoms of a pneumonia:

  * cough which is newly appeared or increasing,
  * dyspnea
  * mucopurulent or purulent sputum,
  * fever (body temperature >= 37.8 degrees Celsius auricalary and/or >= 38,3°C rectal), positive auscultation
* Negative legionella antigen test in the urine
* CRB-65-Index < 3

Exclusion Criteria:

* Hospitalization within the last 28 days (except for the last 72 h)
* Participation in another therapy study within the last 4 weeks with studies admission
* intake of an antibiotic longer than 24 hrs within the last 72 hours before studies admission
* Patients in the pregnancy and nursing phase
* Existence of contraindications opposite the examining preparations or other B-Lactam antibiotics or fluorochinolons
* Patients with a CURB-Index >= 3
* Patients with suspicion of retrostenotic Pneumonia because of bronchial obstruction
* Patients with suspicion of nosocomial Pneumonia
* Patients with an infection by a known or suspected resistant pathogene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2008-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Proof of the clinical non inferiority by the cure rate at the treatment of a Pneumonia at the therapy end (round 3: Day 7 to 10) with a standard penicillin in a high dosage | after at least 7 days, i.e., at the time of round 3 (therapy end)

SECONDARY OUTCOMES:
clinical cure rate | at round 4 (follow-up: day 28 to 35)
bacteriological effectiveness on patients and seed level | at round 4 (follow-up: day 28 to 35)
bacteriological sensitivity into-vitro | at round 4 (follow-up: day 28 to 35)
time up to the drug-switch | at round 4 (follow-up: day 28 to 35)
time until the dismissal of the patients necessity of the gift of additional antibacterial drug | at round 4 (follow-up: day 28 to 35)
cost reduction of the antibiotic-therapy and the complete treatment | at round 4 (follow-up: day 28 to 35)
assessment of the effectiveness by the investigator | at round 4 (follow-up: day 28 to 35)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Welte, Prof., Principal Investigator — Hannover Medical School
Locations (8):
- Germany (8):
  - Charité - Universitätsmedizin Berlin ,Campus Virchow-Klinikum ,Medizinische Klinik : Infektiologie u. Pneumologie, Berlin
  - HELIOS-Klinikum Emil von Behring ,Lungenklinik Heckeshorn, Berlin
  - Klinikum der Ruhr Universität , Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil, Medizinische Klinik III, Bochum
  - Medizinische Hochschule Hannover, Abteilung für Pneumologie, Hanover
  - Universitätsklinikum-Schleswig-Holstein, Campus Lübeck, Zentralklinikum, MK III, Studienzentrum Pneumologie-Infektiologie-Onkologie,, Lübeck
  - Brüderkrankenhaus St. Josef , Innere Abteilung, Paderborn
  - Diakoniekrankenhaus Rotenburg gGmbH, Lungenklinik Unterstedt , Zentrum für Pneumologie, Rotenburg (Wümme)
  - Universitätsklinikum Ulm Sektion Pneumologie/Klinik für Innere Medizin II, Ulm

REFERENCES:
- See also: Related Info — http://www.capnetz.de